CLINICAL TRIAL: NCT07016594
Title: The Effect of Aerobic Exercise With and Without Neuromuscular Electrical Stimulation on Acute Cardiovascular Responses Between Biological Sexes
Brief Title: Acute Cardiovascular Responses to Two Types of Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Stephen Mark Cornish, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HE2021-0209
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Aerobic Exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise alone (Active Comparator): Participants completed aerobic exercise acutely
  Interventions: Behavioral: Aerobic exercise
- Aerobic exercise with neuromuscular electrical stimulation of the leg musculature (Experimental): Participants completed aerobic exercise with neuromuscular electrical stimulation
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — Aerobic exercise was done with and without neuromuscular electrical stimulation

SUMMARY:
The purpose of this research was to explore potential differences in acute cardiovascular responses between two conditions: 1) moderate-intensity cycle ergometer exercise; and 2) moderate-intensity cycle ergometer exercise with NMES. Young, healthy, physically active participants were recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* performing aerobic activity greater than or equal to three times per week at any intensity

Exclusion Criteria:

* had lower body musculoskeletal injuries recently (within the past 6 months)
* health conditions that may place risk to the individual such as those with respiratory issues, hypertension, chronic atrial fibrillation, valvular diseases, heart disease; or obstructive cardiomyopathy
* if taking pharmacological drugs, performance-enhancing drugs, recreational drugs, nutritional supplements, or smoked nicotine

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption | 20 minutes
  L/min

SECONDARY OUTCOMES:
Carbon dioxide production | 20 minutes
  L/min
Heart rate | 20 minutes
  bpm
Respiratory exchange ratio | 20 minutes
  RER (0.70-1.00)
Rating of perceived exertion | 20 minutes
  RPE (6-20)
Kilocalories utilized | 20 minutes
  kcal/min
Carbohydrate utilized | 20 minutes
  g/min
Fats utilized | 20 minutes
  g/min

CONTACTS AND LOCATIONS:
Locations (1):
- Active Living Centre/Applied Research Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Will decide if asked by other investigators.